CLINICAL TRIAL: NCT04840095
Title: Dynamic Connectivity Under Metabolic Constraints
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Martinos Center for Biomedical Imaging (Other)
Responsible Party: Principal Investigator, Lilianne R. Strey, Associate Neuroscientist, Massachusetts General Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 2015P000652
Record Dates: First submitted 2021-04-07; First posted 2021-04-09 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Insulin Resistance; Healthy; Diet Modification; Aging
Keywords: exogenous ketone; insulin resistance; glucose; diet; aging
MeSH Terms: conditions — Insulin Resistance | interventions — Ketones; Glucose

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Metabolic Manipulation via Diet fMRI (Experimental): All subjects are tested three times, each in a different diet-induced metabolic state: glycolytic (glucose burning), fasting (8 hours no food), and ketotic (fat burning). While having their brains scanned with MRI, subjects are initially tested at rest, and then perform a task. Midway through the session, subjects are removed from the scanner and drink up to 75g glucose. Our data analyses quantify network reorganization in response to changing energy constraints (i.e., cognitive demand, fuel).
  Interventions: Drug: Glucose
- Metabolic Manipulation via Ketone Supplement fMRI (Experimental): All subjects are tested twice, both times in a fasting condition (8 hours no food, unrestricted water). While having their brains scanned with MRI, subjects are initially tested at rest, and then perform a task. Midway through the session, subjects are removed from the scanner and drink either of two fuel sources. In the ketotic (ketone burning) session they will drink a ketone sports drink dosed at 395mg/kg. During the glycolytic (glucose burning) session the same subjects will drink a bolus of glucose, calorie-matched to the ketones. Our data analyses quantify network reorganization in response to changing energy constraints (i.e., cognitive demand, fuel).
  Interventions: Drug: Ketones; Drug: Glucose
- Metabolic Manipulation via Ketone Supplement MR/PET (Experimental): All subjects are tested twice, both times in a fasting condition (8 hours no food, unrestricted water). For both sessions, we will intravenously administer the FDG radioisotope continuously throughout the scan. Thus, PET will map glucose uptake across the brain, while we simultaneously use MRS to measure production of the neurotransmitters glutamine and GABA. While having their brains scanned with MR/PET, subjects are initially tested at rest, and then perform a task. Subjects will drink a ketone sports drink dosed at 395mg/kg. During the glycolytic (glucose burning) session the same subjects will drink a bolus of glucose, calorie-matched to the ketones.
  Interventions: Drug: Ketones; Drug: Glucose

INTERVENTIONS:
Drug: Ketones — Sports supplement that is administered mid-scan.
  Arms: Metabolic Manipulation via Ketone Supplement MR/PET; Metabolic Manipulation via Ketone Supplement fMRI
Drug: Glucose — Supplement is administered mid-scan.

SUMMARY:
In this study, we investigate the impact of insulin resistance on the acceleration of brain aging, and test whether increased neuron insulin resistance can be counteracted by utilization of alternate metabolic pathways (e.g., ketones rather than glucose). This study has three Arms, which together provide synergistic data. For all three Arms, subjects are tested in a within-subjects design that consists of 2-3 testing sessions, 1-14 days apart, and counter-balanced for order. During each session we measure the impact of fuel (glucose in one session, ketones in the other) on brain metabolism and associated functioning. For Arms 1-2, our primary experimental measure is functional magnetic resonance imaging (fMRI), which we will use to trace the self-organization of functional networks following changes in energy supply and demand. Arm 1 tests the impact of endogenous ketones produced by switching to a low carbohydrate diet, while Arm 2 tests the impact of exogenous ketones consumed as a nutritional supplement. For Arm 3, we use simultaneous magnetic resonance spectroscopy/positron-emission tomography (MR/PET) to quantify the impact of exogenous ketones on production of glutamate and GABA, key neurotransmitters.

Subjects will be given the option to participate in more than one of the Arms, but doing so is not expected nor required.

Prior to scans, subjects will receive a clinician-administered History and Physical (H&P), which includes vital signs, an oral glucose tolerance test (OGTT), and the comprehensive metabolic blood panel. These will be used to assess diabetes, kidney disease, and electrolytes. If subjects pass screening, they will be provided the option to participate in one or more Arms, which include neuroimaging. To provide a quantitative measure of time-varying metabolic activity throughout the scan, based upon quantitative models of glucose and ketone regulation, as well as to be able to implement safety stopping rules (see below), we will obtain pin-prick blood samples three times: prior to the scan, following consumption of the glucose or ketone drink, and following completion of the scan. To assess effects of increased metabolic demand, we measure brain response to cognitive load, transitioning from resting-state to spatial reasoning through a Tetris task. To assess effects of increased metabolic supply, we measure brain response to glucose or ketone bolus.

ELIGIBILITY:
Exclusion Criteria:

* claustrophobia
* history of neurological disease, heart attack, stroke, kidney disease, or myxedema
* chronic usage of alcohol
* current usage of psychotropic medication
* Type 1 diabetes mellitus
* Regular consumption of insulin, Metformin® or other medications (statins, NSAIDs, beta-blockers, glucocorticoids) that affect glucose and/or insulin utilization.
* difficulty swallowing
* pregnancy
* breastfeeding
* For PET: research imaging-related radiation exposure that exceeds current MGH Radiology Radiation Safety Commitee guidelines.

Inclusion Criteria:

* BMI < 30
* 20/20 vision or correctable to 20/20 with contact lenses
* MRI compatible
* For PET with Optional 150 ml Blood Sampling Only: Must weigh at least 110 lbs to minimize risks per PHRC guidelines.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-06-19 (Actual); Primary Completion 2023-09 (Estimated); Study Completion 2023-09 (Estimated)

PRIMARY OUTCOMES:
fMRI stability measures: endogenous ketones vs exogenous glucose | Within two weeks of enrollment completion
  BOLD signal measurements will be obtained at baseline and during either a glycolytic, fasting, or ketotic state. We hypothesize that ketones provide the brain with greater baseline access to energy, particularly as individuals age and become insulin resistant, and that subsequent ingestion of glucose disrupts this access. We also expect that these effects will become more pronounced when metabolic demands are higher (i.e., task vs resting-state).
fMRI stability measures: exogenous ketones vs exogenous glucose | Within two weeks of enrollment completion
  BOLD signal measurements will be obtained at baseline and following either a glucose or ketone supplement. We hypothesize that ketones provide the brain with greater baseline access to energy, particularly as individuals age and become insulin resistant, and that subsequent ingestion of glucose disrupts this access. We also expect that these effects will become more pronounced when metabolic demands are higher (i.e., task vs resting-state).
PET: glucose uptake and neurotransmitter production with and without ketone supplement | Within two weeks of enrollment completion
  During MR/PET scans, continuous FDG infusion will be used to measure glucose uptake both during rest and task. Magnetic resonance spectroscopy will be used to measure production of neurotransmitters. In individuals who are insulin resistant, we expect to find diminished neurotransmitter levels that will then be replenished through exogenous ketones. We also hypothesize that these effects will become more pronounced when metabolic demands are higher (i.e., task vs resting-state).

SECONDARY OUTCOMES:
Cognitive performance will be assessed and correlated with brain stability values and insulin resistance levels | Within two weeks of enrollment completion

CONTACTS AND LOCATIONS:
Overall Officials: Lilianne Mujica-Parodi, PhD, Principal Investigator — Stony Brook University
Locations (2):
- United States (2):
  - Martinos Center for Biomedical Research, Building 149, Charlestown, Massachusetts
  - Bioengineering Building , Stony Brook University, Stony Brook, New York